CLINICAL TRIAL: NCT04131985
Title: Analgesic Efficacy of Erector Spinae Plane Block for Laparoscopic Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savas Altinsoy, Principal Investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Lap ing Hernia
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Postoperative Pain
Keywords: Laparoscopic inguinal hernia surgery,; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: One group will receive erector spinae plane block, and the other will receive nothing
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spina block (Experimental): After the C7 spinous protrusion is prepared as sterile as T10, the erector spina muscle is seen at the T7 level on the same side as the hernia with the convex probe and block is applied with 0.25% bupivacaine (20 cc).
  All anesthesia procedure will be the same as control group
  Interventions: Procedure: Erector Spina Block
- Control (No Intervention): There were no intervention. All patients will receive pre-oxygenation with O2 100% for 3 min. Anesthesia will be induced by using fentanyl 1-2μg/kg, propofol 2 - 4 mg/kg and rocuronium 0.6 mg/kg will be used for muscle relaxation. Anesthesia will be maintained by controlled ventilation with oxygen and air (50:50) with target of EtCO2≈ 35-40 mmHg. Anesthesia was maintained using remifentanil 0.05-0.1 mcg/kg/min and propofol 80-100 mcg/kg/min via total intravenous micro pump until the surgery was completed. Anesthesia will be discontinued and tracheal extubation will be done once patient fulfilled the extubation criteria.Tramadol 100 mg i.v. will be used before 15 min end of surgery and 20 mL of 25% bupivacaine will be infiltrated to the trochar sites at the end of the surgery. Patient control analgesia device will administer all patients.

INTERVENTIONS:
Procedure: Erector Spina Block — After the C7 spinous protrusion is prepared as sterile as T10, the erector spina muscle is seen at the T7 level on the same side as the hernia with the convex probe and block is applied with 0.25% bupivacaine (20 cc).
  Arms: Erector spina block

SUMMARY:
Postoperative analgesia management in inguinal hernia surgery is difficult because of the content of the surgical procedure. A multimodal approach to postoperative analgesia has recently been proposed. For this reason, various methods are used.Regional blocks, pharmacological treatments are among these methods. Among the regional blocks, ilioinguinal and hypogastric blocks are used more safely and with increasing frequency, especially with the introduction of ultrasonography in the clinic.Forero et al. firstly, erector spinae block which was used for the first time in the treatment of thoracic neuropathic pain has been widely used especially in laparoscopic abdominal surgery and it has taken its place in the literature. It is performed at T4-5 level in breast and thoracic surgery and T7 level in abdominal surgery. In this block, local anesthesia between the erector spina muscle and the transverse protrusion of the vertebra was used to create analgesia in the anterior abdominal wall.

In this study, we planned to investigate degree of postoperative pain, sensory block levels, analgesic consumption, propofol-remifentanyle consumption and side effects of patients undergoing inguinal hernia surgery under general anesthesia with erector spinae block.

DETAILED DESCRIPTION:
Patients in the ASA 1-3 group who underwent laparoscopic inguinal hernia surgery, underwent erector spina block and operated under general anesthesia, will be included in the study. Approximately 50 patients will participate in the study, the number of patients will be finalized by power analysis.

The routine algorithm for patients undergoing elective laparoscopic inguinal hernia surgery is a multimodal approach including induction of general anesthesia for postoperative analgesia followed by peripheral nerve block and 50 mg of dexketoprofen trometamol. Before the block, all patients were monitored by standard monitoring and intravenous vascular access was opened. When applying the erector spinae block, the patient is placed in the lateral decubitus position. After the C7 spinous protrusion is prepared as sterile as T10, the erector spina muscle is seen at the T7 level on the same side as the hernia with the convex probe and block is applied with 0.25% bupivacaine (20 cc). In the control group, there were no intervention except local anesthetic infiltration to the trochar sites. Sensory block was evaluated by cold stimulus (0 = no cold sensation, 1 = cold sensation severely reduced, 2 = cold sensation slightly decreased, 3 = normal cold sensation). In anesthesia induction, propofol 2-4 mg / kg, fentanyl 1-2 mcq / kg, lidocaine 1mg / kg and rocuronium 0.6 mg / kg are routinely administered to all patients. Patients were treated with inhalation of oxygen and air mixture during surgery, and anesthesia was maintained using remifentanil 0.05-0.1 mcg/kg/min and propofol 80-100 mcg/kg/min via total intravenous micro pump until the surgery was completed. Postoperative analgesic needs of the patients will be recorded from the information in the current patient controlled analgesia device. All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Inguinal hernia disease

Exclusion Criteria:

* Cardio-respiratory disease
* Anti-inflammatory treatment
* Cognitive disorders
* Written consent form haven't get
* history of relevant drug allergy
* infection of the skin at the site of needle puncture area
* coagulopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
The degree of postoperative pain | 1hour
  The degree of pain will be measured with numerical rating scale (NRS). All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.
The degree of postoperative pain | 6 hours after operation
  The degree of pain will be measured with numerical rating scale (NRS). All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.
The degree of postoperative pain | 12 hours after operation
  The degree of pain will be measured with numerical rating scale (NRS). All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.
The degree of postoperative pain | 24 hours after operation
  The degree of pain will be measured with numerical rating scale (NRS). All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.
The degree of postoperative pain | 0 hour after operation in postanesthesia care unit
  The degree of pain will be measured with numerical rating scale (NRS). All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.
The degree of postoperative pain | 4 hours after operation
  The degree of pain will be measured with numerical rating scale (NRS). All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.

SECONDARY OUTCOMES:
Side effects of opioid usage | 1, 6, 12 and 24 hours after operation
  Any evidence of opioid-related morbidity or adverse effects eg. nausea,vomiting,pruritus.These effects will be assessed by questionnaire as yes or no
Sensory block levels | 1, 6, 12 and 24 hours after operation
  Sensory block will evaluate by cold stimulus (0 = no cold sensation, 1 = cold sensation severely reduced, 2 = cold sensation slightly decreased, 3 = normal cold sensation)
Postoperative tramadol consumption | The first 24 hour after operation
  total tramadol consumption in both groups will be assessed in the postoperative period
Postoperative quality of recovery | One day before surgery in outpatient clinics of anesthesiology, at 6 hours after the operation, and 24 hours after operation
  The quality of postoperative functional recovery was assessed using the QoR-40, which assesses physical comfort (12 items), emotional state (9 items), physical independence (5 items), psychological support (7 items), and pain (7 items). Each item was rated on a 5-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery)

CONTACTS AND LOCATIONS:
Overall Officials: Savas Altinsoy, MD, Principal Investigator — Diskapi Yildirim Beyazit Education and Research Hospital
Locations (1):
- university of health siences diskapi yildirim beyazit T&R hospital, Ankara, Turkey (Türkiye)